CLINICAL TRIAL: NCT03466463
Title: A Phase I/II, Open Label, Study to Evaluate Safety and Efficacy of an Intravenous Injection of GNT0003 (AAV Vector Expressing the UGT1A1 Transgene) in Patients With Severe Crigler-Najjar Syndrome Requiring Phototherapy
Brief Title: Gene Therapy for Severe Crigler Najjar Syndrome
Acronym: CareCN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Genethon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: GNT-012-CRIG
Record Dates: First submitted 2018-02-01; First posted 2018-03-15 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-02

CONDITIONS: Crigler-Najjar Syndrome
Keywords: Crigler-Najjar; Adeno Associated Virus
MeSH Terms: conditions — Crigler-Najjar Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GNT0003 (Experimental): 2 doses of the IMP assessed in the dose escalation, open-label, phase 1/2 study
  Interventions: Genetic: GNT0003

INTERVENTIONS:
Genetic: GNT0003 — Intravenous infusion, single dose

SUMMARY:
This is a Phase 1/2, multinational, open-label, study to evaluate the safety and efficacy of an intravenous infusion of GNT0003 in patients with Crigler-Najjar aged ≥10 years and requiring phototherapy. Patients will received a single administration of GNT0003 and will be followed for safety and efficacy of approximately 60 months (5 years):

* a follow-up of approximately 12 months (48 weeks)
* a long term follow-up of approximately 48 months (4 years), in order to be in line with the latest EMEA Guideline on follow-up of patients administered with gene therapy medicinal products, released on 22 Oct.2009 by the Committee for medicinal products for human use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe Crigler-Najjar syndrome resulting from a molecular confirmation of mutations in the UGT1A1 gene and requiring phototherapy
* Male or female at least 9 years at the date of signature of informed consent
* Patient able to give informed assent and/or consent in writing

Exclusion Criteria:

* Patients who underwent liver transplantation
* Patients with chronic hepatitis B or C
* Patients infected with Human immunodeficiency virus (HIV)
* Patients with significant underlying liver disease
* Patients with significant encephalopathy
* Participation in any other investigational trial during this trial
* Patients unable or unwilling to comply with the protocol requirements

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2030-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients having received the selected dose of GNT0003 with serum bilirubin ≤ 300µmol/L within 48 meeks after GNT0003 administration and without phototherapy from week 16 | 48 weeks
  Decrease of total Serum bilirubin level after interruption of daily phototherapy (Efficacy); change in serum total biliirubin from baseline to week 48
Incidence of Treatment Emergent Adverse Events or Treatement Serious Adverse Events | 48 weeks
  Incidence of AE/SAE evaluated by changes in laboratory parameters, vital signs, physical examination, reported from baseline to each visit study. Clinically relevant abnormal findings on Laboratory values, Vital Signs, Physical findings will be reported as Adverse Events.
  Incidence and Severity of Adverse Events for each body system will be presented for each dose level and summarized overall.

SECONDARY OUTCOMES:
Change in Health-related quality of Life for Adults from Baseline to Week 48 after GNT0003 administration | 48 weeks
  Quality of Life outcome measure: change of quality of life from Baseline to Week 48 after GNT0003 administration.
  Scale 36-Item Short Form Survey (SF-36 Health Survey) for adults: from 0 (negative to health) to 100 (positive to health)
Change in Health-related quality of Life for Children from Baseline to Week 48 after GNT0003 administration | 48 weeks
  Quality of Life outcome measure: change of quality of life from Baseline to Week 48 after GNT0003 administration.
  PedsQL 4.0 Generic Core Scale for pediatrics: 0-100 scale where higher scores indicate better health-related quality of life

CONTACTS AND LOCATIONS:
Overall Officials: LABRUNE Philippe, Prof, Principal Investigator — Hopital Antoine Beclere
Locations (4):
- Hopital Antoine BECLERE, Clamart, France
- Italy (2):
  - ASST Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliera Universitaria Federico II, Napoli
- AMC, Amsterdam, Netherlands

REFERENCES:
- [Derived] D'Antiga L, Beuers U, Ronzitti G, Brunetti-Pierri N, Baumann U, Di Giorgio A, Aronson S, Hubert A, Romano R, Junge N, Bosma P, Bortolussi G, Muro AF, Soumoudronga RF, Veron P, Collaud F, Knuchel-Legendre N, Labrune P, Mingozzi F. Gene Therapy in Patients with the Crigler-Najjar Syndrome. N Engl J Med. 2023 Aug 17;389(7):620-631. doi: 10.1056/NEJMoa2214084. PMID 37585628